CLINICAL TRIAL: NCT07137169
Title: LIMA Protocol Towards Palatal Fistula and Maxillary Growth in Cleft Palate: A Randomized Controlled Trial
Brief Title: LIMA Protocol Towards Palatal Fistula and Maxillary Growth in Cleft Palate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kristaninta Bangun, Principal Investigator, Head of Plastic and Reconstructive Surgery Division, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIMAProtocol
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cleft Palate; Fistula of Soft Palate (Disorder); Maxillar Hypoplasia
Keywords: LIMA Protocol; cleft palate; palatoplasty; cleft palate repair; palatal fistula; maxillary growth restriction
MeSH Terms: conditions — Cleft Palate; Retrognathia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIMA Protocol (Experimental): LIMA Protocol classifies cases of cleft palate based on the cleft severity (using palatal index), and guide which method of cleft palate repair surgery should be done
  Interventions: Procedure: LIMA protocol
- RSCM Protocol (Active Comparator): RSCM Protocol guide which method of cleft palate repair surgery should be done in a cleft palate (without classifying based on cleft palate severity/ palatal index)
  Interventions: Procedure: RSCM Protocol

INTERVENTIONS:
Procedure: LIMA protocol — Cleft palate repair using Hybrid / One-flap technique
  Arms: LIMA Protocol
Procedure: RSCM Protocol — Cleft palate repair using Two-flap technique
  Arms: RSCM Protocol

SUMMARY:
This randomized controlled trial compared palatoplasty outcomes using the LIMA protocol (Hybrid and one-flap techniques) versus the RSCM protocol (two-flap technique) in patients with unilateral Veau III-IV cleft palate at Cipto Mangunkusumo Hospital from January 2022 to December 2024.

DETAILED DESCRIPTION:
Background: Palatoplasty in patients with cleft palate carries risks of palatal fistula and impaired maxillary growth, both of which are influenced by cleft severity and surgical technique. The LIMA protocol offers a refined classification and tailored surgical approach, with promising results in reducing these complications.

Methods: This study is a randomized controlled trial comparing palatoplasty techniques based on the LIMA protocol (Hybrid and one-flap techniques) versus the RSCM protocol (two-flap technique) in terms of surgical outcomes: palatal fistula and maxillary growth. The study was conducted at Cipto Mangunkusumo Hospital (RSCM) from January 2022 to December 2024. Samples were collected consecutively, with all subjects who met the inclusion criteria (patients aged 9 months-2 years with unilateral Veau III-IV cleft palate undergoing primary palatoplasty at RSCM) randomly allocated into two study groups. Data were analyzed using T-test and Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete unilateral cleft lip and palate aged 9 months to 2 years who agreed to be research subjects
* Patients with complete unilateral cleft lip and palate who underwent palatoplasty surgery at Cipto Mangunkusumo Hospital

Exclusion Criteria:

* Patients who refuse to be research subjects and do not want to sign consent form
* Patients with complete unilateral cleft lip and palate who have previously undergone cleft palate repair/ palatoplasty

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Maxillary Size Indicators Observed From Dental Casts | From the time of surgery until 6 months post-operatively
  Maxillary growth is assessed by measuring its size based on indicators obtained from dental casts before surgery, 1 month post-surgery, and 6 months post-surgery.
  There will be 4 indicators, namely:
  1. 'CC = primary inter-canine width
  2. 'TT = inter-tuberosity width
  3. 'ICC = length from incisivus to the 'CC line (indicating anterior palatal length)
  4. 'ITT = length from incisivus to the 'TT line (indicating overall palatal length)
Palatal Fistula by Pittsburgh Classification | From the time of surgery until 6 months post-operatively
  A palatal fistula is an abnormal opening in the palate that persists or develops after cleft palate repair, creating a connection between the oral and nasal cavities, excluding openings due to wound/ suture dehiscence.
  The location of opening will be Classified using Pittsburgh Classification;
  Type I: uvula; Type II: soft palate; Type III: junction between the soft and hard palate; Type IV: hard palate; Type V: junction between the primary and secondary palate; Type VI: lingual-alveolar; Type VII: labial-alveolar.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient privacy and confidentiality, as well as institutional policies that limit the sharing of sensitive clinical data without additional ethical approvals and data use agreements

REFERENCES:
- [Background] Chiu YT, Liao YF. Is cleft severity related to maxillary growth in patients with unilateral cleft lip and palate? Cleft Palate Craniofac J. 2012 Sep;49(5):535-40. doi: 10.1597/10-044. Epub 2010 Dec 23. PMID 21214323
- [Background] Farronato G, Kairyte L, Giannini L, Galbiati G, Maspero C. How various surgical protocols of the unilateral cleft lip and palate influence the facial growth and possible orthodontic problems? Which is the best timing of lip, palate and alveolus repair? literature review. Stomatologija. 2014;16(2):53-60. PMID 25209227
- [Background] Parwaz MA, Sharma RK, Parashar A, Nanda V, Biswas G, Makkar S. Width of cleft palate and postoperative palatal fistula--do they correlate? J Plast Reconstr Aesthet Surg. 2009 Dec;62(12):1559-63. doi: 10.1016/j.bjps.2008.05.048. Epub 2008 Oct 5. PMID 18838320
- [Background] Todorov AB, Bolling DR. A computerized file for studying growth development in achondroplasia. Birth Defects Orig Artic Ser. 1974;10(9):241-4. No abstract available. PMID 4422204
- [Background] Hui BK, Lai LH, Nguyen PD, Yee KS, Martz MG, Bradley JP, et al. Maxillary Hypoplasia in the Cleft Patient: Contribution of Dental Agenesis to Le Fort I Advancement Surgery. Journal of Oral and Maxillofacial Surgery. 2014;72(9):e56-e7.
- [Background] Smith DM, Vecchione L, Jiang S, Ford M, Deleyiannis FW, Haralam MA, Naran S, Worrall CI, Dudas JR, Afifi AM, Marazita ML, Losee JE. The Pittsburgh Fistula Classification System: a standardized scheme for the description of palatal fistulas. Cleft Palate Craniofac J. 2007 Nov;44(6):590-4. doi: 10.1597/06-204.1. PMID 18177198
- [Background] Rossell-Perry P, Caceres Nano E, Gavino-Gutierrez AM. Association between palatal index and cleft palate repair outcomes in patients with complete unilateral cleft lip and palate. JAMA Facial Plast Surg. 2014 May-Jun;16(3):206-10. doi: 10.1001/jamafacial.2013.2537. PMID 24652124
- [Background] Lima Protocol for Cleft Palate Repair in Cleft and Craniofacial Centre Cipto Mangunkusumo Hospital Indonesia: A Preliminary Study. J Plast Rekons. 2024;9(1):7-12.
- [Background] Rossell-Perry P, Cotrina-Rabanal O, Figallo-Hudtwalcker O, Gonzalez-Vereau A. Effect of Relaxing Incisions on the Maxillary Growth after Primary Unilateral Cleft Palate Repair in Mild and Moderate Cases: A Randomized Clinical Trial. Plast Reconstr Surg Glob Open. 2017 Jan 16;5(1):e1201. doi: 10.1097/GOX.0000000000001201. eCollection 2017 Jan. PMID 28203502
- [Background] Rossell-Perry P, Cotrinal-Rabanal O, Caceres-Nano E. One-flap Palatoplasty: A Cohort Study to Evaluate a Technique for Unilateral Cleft Palate Repair. Plast Reconstr Surg Glob Open. 2015 May 7;3(4):e373. doi: 10.1097/GOX.0000000000000342. eCollection 2015 Apr. PMID 25973351
- [Background] Rossell-Perry P, Luque-Tipula M. The Lima Surgical Protocol for Cleft Palate Repair. J Craniofac Surg. 2020 Sep;31(6):1533-1538. doi: 10.1097/SCS.0000000000006331. PMID 32195838
- [Background] Kreshanti P, Sari VA, Wangge G, Wahyuni LK. Speech Outcome Evaluation Of Cleft Palate Patients Underwent Palatoplasty In Plastic Surgery Division Cipto Mangunkusumo Hospital Indonesia. J Plast Rekonst. 2018;5(1):160-70.